CLINICAL TRIAL: NCT04641663
Title: Clinical Trial to Assess Tolerability and Availability of a Multi-target Dietary Supplement in an Aging Population
Brief Title: Multi-target Dietary Supplement Tolerability in an Aging Population (MTDSST)
Acronym: MTDSST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Douglas Boreham (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor-Investigator, Douglas Boreham, Professor/Director - Medical Sciences, Northern Ontario School of Medicine
Organization: Northern Ontario School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTDS-001
Record Dates: First submitted 2020-11-12; First posted 2020-11-24 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Aging; Age-related Cognitive Decline
Keywords: Dietary Supplement; Aging; Safety; Tolerability

STUDY DESIGN:
Intervention Model Description: participants will be taking either 60%, 80% or 100% of the recommended daily dose of the dietary supplement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100 RDD (Experimental): 100% of recommended daily dose (RDD) of the MORNING tablet dose (5 tablets), all groups will receive the full recommended dose for both EVENING (3 tablets) and OMEGA (2 softgels) doses.
  Interventions: Dietary Supplement: Multi-target Dietary Supplement (MTDS)
- 80 RDD (Experimental): 80% of recommended daily dose of the MORNING tablet dose (4 tablets), all groups will receive the full recommended dose for both EVENING (3 tablets) and OMEGA (2 softgels) doses.
  Interventions: Dietary Supplement: Multi-target Dietary Supplement (MTDS)
- 60 RDD (Experimental): 60% of recommended daily dose of the MORNING tablet dose (3 tablets), all groups will receive the full recommended dose for both EVENING (3 tablets) and OMEGA (2 softgels) doses.
  Interventions: Dietary Supplement: Multi-target Dietary Supplement (MTDS)

INTERVENTIONS:
Dietary Supplement: Multi-target Dietary Supplement (MTDS) — The Multi-Target Dietary Supplement (MTDS) is comprised of 51 ingredients designed to simultaneously target and support the cellular processes implicated in the progression of the aging phenotype (oxidative stress, inflammatory processes, insulin resistance, and membrane and mitochondrial deterioration). The MTDS is unique in that it was specifically designed as a multi-target intervention to support the complex cellular perturbations associated with aging. Components of the formulation were chosen based on scientific consensus of documented effectiveness for one or more of the targeted processes, long-term evidence of safety, and synergistic or additive interactions between components.
  The MTDS is divided into morning and evening doses to maximize availability of the components to the peak activity level of the cellular processes that require those components.
  Other Names: AS-10 Plus

SUMMARY:
This study is being performed to determine if a multi-ingredient dietary supplement is safe and easy to take by healthy older adults. Participants will be required to take one of three different doses of the dietary supplement for 90 consecutive days and complete wellness surveys and a daily log while taking the supplement. Participants will also provide blood samples at the start of the study, after 30 days, and at the end of the study which will help determine how participants respond to the supplement.

DETAILED DESCRIPTION:
Likely because of the highly complex nature of aging, there has been little success reducing age-related physical and cognitive deterioration. The predominant approach has been to manage emergent symptoms rather than mitigate the cellular mechanisms driving the degenerative processes underlying aging. Additionally, the multifaceted and complex etiology of aging makes it extremely difficult to provide effective interventions within current treatment paradigms. The medical community has established that preventative measures are the most effective means of slowing the progression of age-associated deterioration, however effective methods or interventions have not been established.

The Multi-Target Dietary Supplement (MTDS) was designed to simultaneously target and support the cellular processes implicated in the progression of the aging phenotype (oxidative stress, inflammatory processes, insulin resistance, and membrane and mitochondrial deterioration). The MTDS is unique in that it was specifically designed as a multi-target intervention to support the complex cellular perturbations associated with aging. Components of the formulation were chosen based on scientific consensus of documented effectiveness for one or more of the targeted processes, long-term evidence of safety, and synergistic or additive interactions between components.

In more than 20 years of pre-clinical research, the MTDS has demonstrated significant beneficial impacts in animal models of aging and age-associated disease. The MTDS has resulted in significant reductions in both acute and chronic oxidative stress, greatly improved mitochondrial function and efficiency, significantly reduced inflammatory processes and improved glucose metabolism. Signal transduction is normalized to youthful levels in aged animals, including key pathways implicated in aging (unpublished data). On a functional level, MTDS treatment has resulted in increased longevity of 10 to 28% in normal and accelerated aging phenotypes, respectively. Concomitant improvements in mobility, activity levels, muscle strength (exercise mimetic) and overall body condition in aged animals were observed. Dramatic reductions in the incidence of muscle wasting, arthritic processes, and cataracts were also observed. Sensory and cognitive acuity were protected and frequently enhanced in aged animals, with significant improvements in visual and olfactory function observed in a broad range of tasks. MTDS treatment has demonstrated profound sparing from age-related neuronal losses and corresponding protection of neurogenesis and enhanced synaptogenesis, resulting in dramatically improved cognition in aged animals. The quantity of data indicating MTDS efficacy in pre-clinical studies is considerable, however the effects of the MTDS in humans, although positive, remains anecdotal. This tolerability study is the critical first step to begin assessment of the efficacy of the MTDS in human populations. If even a portion of these protective effects of the MTDS are translatable from mice to humans, the positive impacts for the aging population and Ontario's healthcare system could be profound.

This is a multi-center, three-arm study designed to evaluate the safety of a dietary supplement at three dosing regimes for 90 days. Initially, 45 healthy volunteers will be randomly assigned to one of three dose regimes: 1) 100% of recommended daily dose (RDD), 2) 80% of recommended daily dose or 3) 60% of recommended daily dose. Dosing regimes are based on levels of the MORNING tablet doses, all groups will receive the full recommended dose for both EVENING and OMEGA doses. Written informed consent will be obtained and a medical history and health assessment will be performed. The investigator will determine whether the subject meets all inclusion and exclusion criteria. Health assessments will be made at baseline, 30 days and 90 days. Adverse events, concomitant medications, and product administration will be recorded throughout the study.

Compliance, safety, and tolerability parameters are the primary focus of this study; however the probability of serious adverse events is extremely low given the long safety history of safety of the vitamins and nutraceuticals that comprise the MTDS.

The primary objective is to evaluate the safety and tolerability of the MTDS regimen in terms of its administration at 3 dosing regimes for 90 consecutive days with respect to micronutrient levels, laboratory tests and adverse events.

The secondary objectives include:

1. monitoring compliance of taking the MTDS,
2. monitoring wellness as measured by the 36-Item Short Form Survey (SF-36) scale and daily journal, over the 90-day administration of the MTDS, and
3. to assess MTDS absorption through plasma micronutrient testing, at baseline, 30 days and 90 days following administration of the test agent.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects ages of 45 and older.
2. Capable of providing informed consent
3. Patients currently taking fluconazole, 3-hydroxy-3-methyl-glutaryl-CoA reductase (HMG-CoA) reductase inhibitors (i.e. "statin" drugs), or any other drug known to interfere with serum transaminase (i.e. liver enzymes), must have history of stable liver function test since first taking such drugs.
4. Patients who usually and customarily take dietary supplements, including vitamins, must undergo a two-week washout period

Exclusion Criteria:

1. Exposure to any investigational drug within 90 days of the beginning of this study
2. Known human immunodeficiency virus (HIV) seropositivity or Acquired Immunodeficiency Syndrome (AIDS); history of Hepatitis B (HBV), Hepatitis C (HCV) vital infection, unexplained elevated serum transaminase, or other hepatic disease. NOTE: HIV, HCV, and HBV testing will not be performed as part of screening.
3. History of cancer within the last 5 years, except for basal or squamous cell cancer.
4. Recent COVID-19 infection.
5. Allergy to fish (specifically sardines, anchovies or mackerel) or any of the investigational product components
6. Concomitant use, or use within less than a two-week period, of any other dietary supplement
7. Concomitant use of any drug known to interfere with laboratory measures such as:

   1. Niaspan (extended release niacin)
   2. Lamisil (terbinafine HCl)
   3. Chronic use of acetaminophen (>1,500 mg/day) (occasional use for minor aches and pains is excluded from this restriction)
   4. Newly prescribed (< 90days) HMG-CoA reductase inhibitors ("statin medications"), or patients currently on statin medications who have previously shown evidence of elevated serum transaminases
8. Currently diagnosed with multiple sclerosis, systemic lupus erythematosis, or other autoimmune disorders known to interfere with laboratory measures
9. History of alcoholism or drug abuse, unless it is determined that such past use would not influence laboratory measures (DSN4 criteria)
10. Any other active disease of a life-threatening nature or laboratory abnormality that, in the judgment of the investigator, may interfere with the interpretation, or increase risk of patient participation
11. Conditions that require nutritional therapy, such as:

    1. Pernicious anemia
    2. Iron-deficiency anemia
    3. Hartnup Disease or Pellagra
    4. Scurvy
    5. Beriberi-induced Endemic Neuritis

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2023-09-21 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events (AE) as Assessed by CTCAE v5.0 | out to 90 days
  Subjects are instructed to log any AEs that occur at any time during the study in the study journal. Participants will be contacted by phone after 7 days on the MTDS to assess any occurrence of AEs. Reported or observed AEs will be documented and followed to resolution.
Hematocrit (%) | out to 90 days
  Safety Assessment in Hematology
Hemoglobin (g/L) | out to 90 days
  Safety Assessment in Hematology
Erythrocytes (10^12/L) | out to 90 days
  Safety Assessment in Hematology
Leukocytes (10^9/L) | out to 90 days
  Safety Assessment in Hematology
Basophils (10^3/uL) | out to 90 days
  Safety Assessment in Hematology
Basophils/Leukocytes (%) | out to 90 days
  Safety Assessment in Hematology
Eosinophils (10^9/L) | out to 90 days
  Safety Assessment in Hematology
Eosinophils/Leukocytes (%) | out to 90 days
  Safety Assessment in Hematology
Lymphocytes (10^9/L) | out to 90 days
  Safety Assessment in Hematology
Lymphocytes/Leukocytes (%) | out to 90 days
  Safety Assessment in Hematology
Monocytes (10^9/L) | out to 90 days
  Safety Assessment in Hematology
Monocytes/Leukocytes (%) | out to 90 days
  Safety Assessment in Hematology
Neutrophils (10^9/L) | out to 90 days
  Safety Assessment in Hematology
Neutrophils/Leukocytes (%) | out to 90 days
  Safety Assessment in Hematology
Platelet Count (10^9/L) | out to 90 days
  Safety Assessment in Hematology
Serum Glucose (mmol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Sodium (mmol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Potassium (mmol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Calcium (mmol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Chloride (mmol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Urea (mmol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Creatinine (umol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Urate (umol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Albumin (g/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Alkaline Phosphatase (U/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Aspartate Phosphatase (U/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Alanine Transaminase (U/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Gamma Glutamyl Transpeptidase (U/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Total Bilirubin (umol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Direct Bilirubin (umol/L) | out to 90 days
  Safety Assessment in Serum Chemistry
Lactate Dehydrogenase (U/L) | out to 90 days
  Safety Assessment in Serum Chemistry
High Sensitivity C-Reactive Protein (mg/L) | out to 90 days
  Safety Assessment in Serum Chemistry

SECONDARY OUTCOMES:
Vitamin A (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin B1 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin B2 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin B3 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin B6 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin B12 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Biotin (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Folate (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Pantothenate (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin C (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin D3 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Vitamin K2 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Magnesium (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Manganese (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Zinc (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Copper (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Alpha Lipoic Acid (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Glutamine (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Glutathione (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Carnitine (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Choline (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Inositol (mg/L) | out to 90 days
  Plasma Micronutrient Levels
Coenzyme Q10 (mg/L) | out to 90 days
  Plasma Micronutrient Levels
36-Item Short Form Survey (SF-36) | up to 90 days
  The SF-36 wellness questionnaire will be used to assess the health status of subjects. There are 36 individual questions which identify eight different facets of wellness. These have been described as physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These facets are further collapsed into physical and mental component summaries. The eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This questionnaire will be included in the study booklet given to each subject, and will be self administered.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Boreham, PhD, Principal Investigator — Northern Ontario School of Medicine
Locations (2):
- Canada (2):
  - Northern Ontario School of Medicine - Elliot Lake site, Elliot Lake, Ontario
  - McMaster University - Behavioural Neurosciences, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers outside the study team.